CLINICAL TRIAL: NCT06713993
Title: Noninvasive Testing Procedures, Role of Biomarkers and Anticancer Treatments in Esophageal and Esophagogastric Cancer Survival and Quality of Life of Patients With Cancer of the Esophageopharyngeal and Oesophageophageophageal Junction
Brief Title: Semmelweis Esophageal Cancer Study: Noninvasive Prognostic Parameters in Patients With Oesophageal and Esophagogastric Junction Cancer
Status: Recruiting | Type: Observational
Sponsor: Semmelweis University (Other)
Responsible Party: Sponsor
Other Study IDs: NNGYK/18646-5/2024
Record Dates: First submitted 2024-10-09; First posted 2024-12-03 (Actual); Last update posted 2024-12-03 (Actual); Status verified 2024-09

CONDITIONS: Esophageal Cancer (EsC)
Keywords: Esophageal cancer; heart failure; sarcopenia; malnutrition; frailty; heart function; Esophageal cancer surgery; cardiovascular abnormalities
MeSH Terms: conditions — Esophageal Neoplasms; Heart Failure; Sarcopenia; Malnutrition; Frailty; Cardiovascular Abnormalities

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — Frozen tissue, fixed tissue
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The objective of this observational study was to gain a deeper understanding of the epidemiology of the disease in Hungary through a broad analysis of patients with new-onset esophageal-oesophageal-stomach junction tumors, and to identify key parameters that could potentially influence the outcome of the disease and are closely correlated with morbidity and mortality. The investigators' primary objective is to identify potential factors and conditions that could be influenced and modified to enhance the disease outcome.

Main questions:

1. What are the measurable changes in performance, workload, nutritional status, cardiac function, mental status in the patients studied?
2. What is the time course of the changes during and after treatment?
3. Which pathological parameters are associated with disease outcome and which are potential points of intervention to improve the course of the disease?

Patients will undergo a detailed physical and nutritional assessment, non-invasive imaging tests and several questionnaires in addition to the usual pre- and post-operative examinations.

DETAILED DESCRIPTION:
Detailed assessment of the baseline cardiovascular risk and status (anthropometric data, physical status assessment, psychological and quality-of-life questionnaire, questionnaires on morbidity and cancer-related fatigue, 12-lead ECG, laboratory parameters, body composition, coronary CT, echocardiography and cardiac MR scan).

In addition to the conventional echocardiographic and cardiac MR parameters, the investigators also aimed to determine myocardial deformation, i.e. strain (Medis Suite QStrain) and T1 and T2 mapping values and late-type contrast enhancement and to investigate their prognostic role. To determine late-type contrast accumulation and to determine ECV (extracellular volume), patients will be given Gadovis contrast media.

At the same time as the cardiac MR scan (V0 and V4), a serum blood sample will be taken from the patients, from which the markers below will be measured. These markers are proteins or molecules that potentially play an important role in the development of tumour cachexia. The investigators aim to determine the prognostic significance of these parameters. (Myostatin, IGF-1 (Insulin-like Growth Factor 1), GDF-15 (Growth Differentiation Factor 15), IL-6 (Interleukin-6).

Patients are followed up for cardiovascular complications during anti-tumour treatment and are taken into care.

Patients will be assessed at first presentation, after neoadjuvant treatment, immediately before surgery, in the third week after surgery and in the 3rd, 6th, 9th, 12th postoperative months. Further follow-up is done by outpatient examination, by telephone or e-mail and through the eHealth system of Hungary (EESZT) until the end of the 3rd year.

Patient education:

The detailed patient information leaflet was prepared by the doctors involved in the development of the protocol at Semmelweis University.

Data storage and data protection:

Patients enrolled in the study will be given a unique identifier after enrolment. Only this unique identifier will be used in the research record, so the record will not be directly linked to the patient. No unique identifier (name, place and date of birth, clinical triage number, social security number, ID card number, etc.) will be included in the research form. A separate, locked document will be used to link the unique identifier to the patient. The system-generated unique identifier code is recorded by the clinician on paper, complete with name, social security number and patient´s social security number, prior to the first data entry. The same document contains the patient´s informed consent for the use of the data for scientific purposes. The database and the information and consent forms, including the patient´s signature, are stored by the institute coordinators.

Statistical methods:

Using TIBCO Statistica™ 13.4 software, the normality of continuous variables is tested using the Kolmogorov-Szmirnov test. A two-sample t-test is used for normal distribution assuming a two-tailed distribution and a one-tailed distribution for selected variables (Mandard Score for tumour regression). For variables with non-normal distribution, a Mann-Whitney U test is used as a non-parametric test. Long-term survival data are analysed using Kaplan-Meyer analysis and log rank test.The level of significance is set at p<0.05

Ethical requirements

The research design was drawn up in accordance with current legislation and the World Medical Assotiation´s Declaration of Helsinki.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18 years
* Diagnosis of new-onset esophageal, esophagogastric junction tumor
* Elective curative surgery (open/laparoscopic regardless of surgical technique)
* Patients who have not yet received oncological treatment for their present disease

Exclusion Criteria:

* Lack of consent
* Lack of cooperation
* Contraindications for some studies: If MR scan is contraindicated, cardiac MR scan is not performed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with primary operable oesophageal and oesophagogastric junction tumours presenting to the upper gastrointestinal outpatient clinic at Semmelweis University.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-09-10 (Actual); Primary Completion 2029-09-30 (Estimated); Study Completion 2034-09-10 (Estimated)

PRIMARY OUTCOMES:
Changes in cardiac function: cardiac MR scan | From enrollment to the 12th postoperative month
  Assessment of cardiac function by cardiac MR scan before starting treatment, after surgery and at postoperative month 12.
Changes in coronary status: coronary CT scan | From enrollment to the 12th postoperative month
  Assessment of coronary status by coronary CT scan before starting treatment, after surgery and at postoperative month 12.
Morbidity (early and long term) classified after Clavien-Dindo. | 30 days (until 31st postoperative day)
  7-day and 30-day morbidity will be detailed assessed. Grade 3 or above morbidity rate will be assessed.
Early and late mortality | 90 days (until 91st postoperative day)
  7-day, 30-day and 90-day mortality of each patient will be recorded
Length of hospital stay | within 45 days
  Postoperative length of hospital stay in days.
Number of days spent on ICU (Intensive care unit) | within 45 days postoperative
  Number of days observed on ICU right after operation.
Changes in physical performance: 6-minute walk test (6MWT) | From enrollment to the 12th postoperative month
  6-minute walk test (6MWT) assessment at the first appointment, immediately before surgery, third week postoperatively and postoperative 3. 6. 9. 12. months.
Changes in physical performance: hand grip strength test | From enrollment to the 12th postoperative month
  Hand grip strength test assessment at the first appointment, immediately before surgery, third week postoperatively and postoperative 3. 6. 9. 12. months.
Changes in physical performance: time up and go test | From enrollment to the 12th postoperative month
  Time up and go test assessment at the first appointment, immediately before surgery, third week postoperatively and postoperative 3. 6. 9. 12. months.
Changes in ECOG (Eastern Cooperative Oncology Group) performance status | From enrollment to the 12th postoperative month
  ECOG (Eastern Cooperative Oncology Group) performance status assessment at the first appointment, immediately before surgery, third week postoperatively and postoperative 3. 6. 9. 12. months.
Change in nutritional status, risk of malnutrition and nutritional ability: MUST (Malnutrition Universal Screening Tool) | From enrollment to the 12th postoperative month
  Malnutrition Universal Screening Tool (MUST) score recording at the first encounter, immediately before surgery, third week post-operatively and post-operatively 3. 6. 9. 12. months. 0-2: If a patient receives a score of 0, then they are at a low risk. A patient with a score of 1 is a medium risk and any patient with a score of 2 or higher is considered high risk.
Change in nutritional status, risk of malnutrition and nutritional ability: NRS (nutritional risk score) | From enrollment to the 12th postoperative month
  NRS (nutritional risk score) recording at the first encounter, immediately before surgery, third week post-operatively and post-operatively 3. 6. 9. 12. months.
  From enrollment to the 12th postoperative month Score 0-3: 0: absent, 3: severe
Change in nutritional status, risk of malnutrition and nutritional ability Description: PG-SGA (Patient-Generated Subjective Global Assessment)score | From enrollment to the 12th postoperative month
  PG-SGA (Patient-Generated Subjective Global Assessment) score recording at the first encounter, immediately before surgery, third week post-operatively and post-operatively 3. 6. 9. 12. months. The PG-SGA allows to classify nutritional status into three categories: A= well nourished; B= suspected or moderate malnutrition; and C= severe malnutrition.
Change in nutritional status, risk of malnutrition: Bioimpedance examination | From enrollment to the 12th postoperative month
  Bioimpedance examination recording at the first encounter, immediately before surgery, third week post-operatively and post-operatively 3. 6. 9. 12. months.
Change in nutritional ability: swallowing test | From enrollment to the 12th postoperative month
  Swallowing test recording at the first encounter, immediately before surgery, third week post-operatively and post-operatively 3. 6. 9. 12. months.
Change in nutritional status: myostatin level | From enrollment to the 12th postoperative month
  Measurement of myostatin level before the start of treatment, postoperatively and at postoperative month 12.
Change in nutritional status: IGF-1 level | From enrollment to the 12th postoperative month
  Measurement of serum IGF-1 level before the start of treatment, postoperatively and at postoperative month 12.
Change in nutritional status: GDF-15 level | From enrollment to the 12th postoperative month
  Measurement of serum GDF-15 level before the start of treatment, postoperatively and at postoperative month 12.
Change in nutritional status: IL-6 level | From enrollment to the 12th postoperative month
  Measurement of serum IL-6 level before the start of treatment, postoperatively and at postoperative month 12.

SECONDARY OUTCOMES:
Change in mental status: adherence | From enrollment to the 12th postoperative month
  Completion of MAS-12 (Motivation Assessment Scale) questionnaire at first appointment, immediately before surgery, third week post-operatively and post-operatively 3. 6. 9. 12. months The MAS-12 total score ranges from 12 to 60 (higher score indicates higher treatment adherence)
Change in cancer related fatigue | From enrollment to the 12th postoperative month
  Brief Fatigue Inventory (BFI) questionnaires at first appointment, immediately before surgery, third week post-operatively and post-operatively 3. 6. 9. 12. months Scoring respondents rate each item on a 0-10 numeric scale, with 0 meaning "no fatigue" and 10 meaning "fatigue as bad as you can imagine." Scores are divided into 3 categories based on the average of each response categorized as mild (1-3), moderate (4-6), and severe (7-10).
Delay in beginning of adjuvant oncotherapy (chemotherapy, radiotherapy). | within 8 weeks, if adjuvant oncotherapy is needed
  Sufficient recovery time until fitness of adjuvant chemo/radiotherapy will be recorded.
Change in mental status: depression | From enrollment to the 12th postoperative month
  Completion of PHQ-9 (Patient Health Questionnaire-9) questionnaire at first appointment, immediately before surgery, third week post-operatively and post-operatively 3. 6. 9. 12. months The PHQ-9 total score ranges from 0 to 27 (scores of 5-9 are classified as mild depression; 10-14 as moderate depression; 15-19 as moderately severe depression; ≥ 20 as severe depression)
Change in mental status: anxiety | From enrollment to the 12th postoperative month
  GAD-7 (General Anxiety Disorder) questionnaire at first appointment, immediately before surgery, third week post-operatively and post-operatively 3. 6. 9. 12. months GAD-7 total score for the seven items ranges from 0 to 21. 0-4: minimal anxiety. 5-9: mild anxiety. 10-14: moderate anxiety. 15-21: severe anxiety.
Change in frailty: Clinical frailty scale (CFS) | From enrollment to the 12th postoperative month
  Clinical frailty scale (CFS) questionnaire at first appointment, immediately before surgery, third week post-operatively and post-operatively 3. 6. 9. 12. months The clinical frailty scale is a 9-point scale that quantifies frailty based on function in individual patients. It is complemented by a visual chart to assist with the classification of frailty. Higher scores indicate increased frailty and associated risks.
Change in frailty: FRAIL scale | From enrollment to the 12th postoperative month
  FRAIL (Fatigue, Resistance, Ambulation, Illness, and Loss) scale questionnaire at first appointment, immediately before surgery, third week post-operatively and post-operatively 3. 6. 9. 12. months The FRAIL scale includes 5 components: Fatigue, Resistance, Ambulation, Illness, and Loss of weight (10). Frail scale scores range from 0-5 (i.e., 1 point for each component; 0=best to 5=worst) and represent frail (3-5), pre-frail (1-2), and robust (0) health status.
Change in frailty: 5-item Frailty Score | From enrollment to the 12th postoperative month
  5-item Frailty Score questionnaire at first appointment, immediately before surgery, third week post-operatively and post-operatively 3. 6. 9. 12. months Scored from 0 to 5 Higher number indicates higher frailty

CONTACTS AND LOCATIONS:
Locations (1):
- Semmelweis University, Budapest, Hungary

IPD SHARING:
Plan to Share IPD: Yes
IPD used in the results publication
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Starting 6 months after publication
Access Criteria: Access to the data is available to any researcher who wishes to use the results for further research (e.g. meta-analysis, sytematic review). The request must be submitted to the research coordinator in the form of a formal e-mail. Data will be provided electronically after a data sharing agreement has been signed. The statistical methods for the analyses and the results must be approved by independent review.

REFERENCES:
- [Background] Lorusso A, Bichev D, Hogner A, Bartels P, Ballhausen A, Treese C, Biebl M, Thuss-Patience P. Prognostic Relevance of Weight and Weight Loss during Multimodal Therapy for Oesophagogastric Tumours. Curr Oncol. 2022 Apr 12;29(4):2706-2719. doi: 10.3390/curroncol29040221. PMID 35448195
- [Background] van Hagen P, Hulshof MC, van Lanschot JJ, Steyerberg EW, van Berge Henegouwen MI, Wijnhoven BP, Richel DJ, Nieuwenhuijzen GA, Hospers GA, Bonenkamp JJ, Cuesta MA, Blaisse RJ, Busch OR, ten Kate FJ, Creemers GJ, Punt CJ, Plukker JT, Verheul HM, Spillenaar Bilgen EJ, van Dekken H, van der Sangen MJ, Rozema T, Biermann K, Beukema JC, Piet AH, van Rij CM, Reinders JG, Tilanus HW, van der Gaast A; CROSS Group. Preoperative chemoradiotherapy for esophageal or junctional cancer. N Engl J Med. 2012 May 31;366(22):2074-84. doi: 10.1056/NEJMoa1112088. PMID 22646630
- [Background] Sondergaard MMA, Nordsmark M, Nielsen KM, Poulsen SH. Cardiovascular Burden and Adverse Events in Patients With Esophageal Cancer Treated With Chemoradiation for Curative Intent. JACC CardioOncol. 2021 Dec 21;3(5):711-721. doi: 10.1016/j.jaccao.2021.10.002. eCollection 2021 Dec. PMID 34988480
- [Background] Eads JR. Cardiovascular Concerns in the Management of Esophageal Cancer Patients. JACC CardioOncol. 2021 Dec 21;3(5):722-724. doi: 10.1016/j.jaccao.2021.11.005. eCollection 2021 Dec. PMID 34988481